CLINICAL TRIAL: NCT06770413
Title: Diagnostic Value of Modified Cough Reflex Test With Staged Water Swallow Test in Post-Stroke Patients Showing Dysphagia
Status: Completed | Type: Observational
Sponsor: Yonsei University (Other)
Responsible Party: Sponsor
Other Study IDs: 4-2019-0111
Record Dates: First submitted 2025-01-07; First posted 2025-01-13 (Actual); Last update posted 2025-01-13 (Actual); Status verified 2025-01

CONDITIONS: Stroke; Pneumonia; Aspiration; Deglutition Disorders
MeSH Terms: conditions — Stroke; Pneumonia; Deglutition Disorders

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Pneumonia group: stroke patients who were diagnosed with pnuemonia within 4 week follow up period
- non-Pneumonia group: stroke patients who were not diagnosed with pnuemonia within 4 week follow up period

SUMMARY:
The investigators conducted staged water swallow test (sWST) and modified cough reflex test (mCRT) on stroke patients referred for videofluoroscopic swallowing studies (VFSS) due to dysphagia. The patients were followed for up to four weeks to examine the incidence and timing of aspiration pneumonia, the relationship between these tests and VFSS results, and the diagnostic value of these tests as screening tools. Descriptive statistics will be presented for the incidence and timing of pneumonia, as well as the results of the SWST and MCRT. Regression analysis will be conducted to determine the explanatory power of each aspiration indicator (sWST and mCRT) in predicting aspiration or aspiration pneumonia. Additionally, using the VFSS results and the diagnosis of aspiration pneumonia as gold standards, the validity, sensitivity, specificity, positive predictive value (PPV), negative predictive value (NPV), odds ratio (OR), and relative risk (RR) for sWST, mCRT, and their combination will be calculated to evaluate their diagnostic value.

ELIGIBILITY:
Inclusion Criteria:

* either ischemic or hemorrhagic stroke confirmed by a computed topography or magnetic resonance imaging
* aged 20 years or older
* signs or symptoms of dysphagia.

Exclusion Criteria:

* inability to maintain sitting posture with support
* dyspnea requiring oxygen supplementation
* diagnosed with aspiration pneumonia at enrollment
* diagnosed with co-existing major neuromuscular disorders affecting swallowing
* diagnosed with infectious diseases requiring isolation
* refusal to participate

Ages: 20 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Stroke patients who were admittied to a single tertiary hospital and demonstrating signs of dysphagia. Dysphagia was documented when any of the following criteria were met: impaired sensory or motor function of oral cavity structures (jaw, lip, tongue, palate, and cheeks), impaired cranial nerve functions (trigeminal, facial, glossopharyngeal, and hypoglossal nerves), voice change (wet or gurgly voice) after swallowing, drooling, or buccofacial apraxia.
Sampling Method: Non-Probability Sample
Enrollment: 328 (Actual)
Dates: Start 2019-05-07 (Actual); Primary Completion 2024-02-28 (Actual); Study Completion 2024-02-28 (Actual)

PRIMARY OUTCOMES:
Incidence of pnuemonia | within 4 weeks after initial evaluation
  Pneumonia was diagnosed using the Mann criteria (when three or more of the following criteria were met: fever (>38°C), productive cough with purulent sputum, abnormal respiratory examination (tachypnea >22/min, tachycardia, inspiratory crackle, bronchial breathing), abnormal chest radiographic findings, arterial hypoxemia (PO2 <70mmHg or SpO2 <94%), and isolation of a relevant pathogen (positive gram stain or culture))

CONTACTS AND LOCATIONS:
Locations (1):
- Severance hospital, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: Undecided
Individual participant date that uderlie the results reported in this article, after deidentification. Study protocol, statistical analysis plan will also be available. Data will be available to researchers who provide a methodologically sound proposal. Proposals should be directed to kimdy@yuhs.ac